



## PERCUTANEOUS ELECTRICAL NERVE STIMULATION OF THE MANDIBULAR NERVE FOR THE MANAGEMENT OF PAIN AND FUNCTIONALITY IN PATIENTS WITH TEMPOROMANDIBULAR DISORDERS.

| Controlled and Randomized Trial. | | | |
|---|---|---|---|
| INFORMED CONS | ENT | | |
| Me : | | | |
| that I have understoo<br>ask the questions the<br>express my free and<br>and I hereby acknow | od what it puts in it<br>at I have considered<br>informed will to vol<br>vledge and agree tha<br>by my signature, to | and that I h<br>necessary<br>luntarily aco<br>at a copy o<br>the proces | at has been handed to me. I affirm have been given the opportunity to in order to understand it well, so I dept my participation in the study, of this consent is given to me and I dissing of my personal data for the desearch project. |
| Place: | Date: | of | 20 |
| Name and surname | of the participant//r | epresentati | ive: |
| Name and surname | of the/the researche | er/: | |
| Signature of the participant | | | Signature of the researcher |



## RIGHT OF REVOCATION (If you wish to exercise your right to withdraw your consent) Me, (name/participant/patient or representative as appropriate): On behalf of myself/or (tick as appropriate) I revoke the informed consent granted to day ...... of ......., no wishing to continue with the study and to terminate it from the date described above. In addition, I agree that a copy of this revocation is given to me. Name and surname of the participant/representative: Name and surname of the/the researcher/: Signature Signature

DATE: 25/7/2023 NCT: 2006202325523